CLINICAL TRIAL: NCT05788250
Title: Randomized Clinical Trial Comparing Rotator Cuff Repair (RCR) With Subacromial Balloon Spacer (SBS) Implantation
Brief Title: RC Repair Versus Subacromial Balloon Spacer in Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Panam Clinic (Other)
Collaborators: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCBAL-01-2023
Record Dates: First submitted 2023-02-01; First posted 2023-03-28 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-04

CONDITIONS: Rotator Cuff Tears
Keywords: rotator cuff repair; subacromial spacer; older adults
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Intervention Model Description: This a double-blind (patient and assessor), parallel, 1:1 multicentre randomized pilot study comparing patients 70 years and older randomized to SBS or RCR. 32 participants from eight orthopaedic surgeons at four sites will be recruited over a one-year period. Randomization will be generated using a web-based system pre-operatively and stratified to ensure 8 medium/large tears and 8 massive tears are allocated to each group.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be blinded to their group allocation. This is possible because the incision and rehabilitation processes are consistent between groups. It is not possible for the treating surgeon to be blinded to group allocation, therefore a research team member (athletic or physical therapist) will remain blinded to group allocation and conduct all study related assessments as well as administer the patient-reported questionnaires. This will be maintained by the participant not removing their shirt during the study assessment. Patients will not be informed of which procedure they will undergo until the study is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subacromial spacer implantation (Experimental)
  Interventions: Procedure: Subacromial spacer implantation
- Rotator Cuff Repair (Active Comparator)
  Interventions: Procedure: Rotator cuff repair

INTERVENTIONS:
Procedure: Subacromial spacer implantation — A biodegradable balloon implanted arthroscopically between the acromion and humeral head with tenotomy of long head of biceps.
  Arms: Subacromial spacer implantation
Procedure: Rotator cuff repair — Rotator cuff repair with tenotomy of long head of biceps.
  Arms: Rotator Cuff Repair

SUMMARY:
The purpose of this pilot study is to assess the feasibility of a full randomized trial design.

DETAILED DESCRIPTION:
The feasibility objectives are:

1. Recruitment

   1. To establish an estimate of the proportion of patients screened who are eligible for inclusion, and of those, the proportion who consent.
   2. To establish an estimate of the proportion of eligible patients with medium/large tears versus massive tears.
2. Surgery -to confirm agreement among surgeons regarding the protocol's standardized surgical techniques of both groups.

Clinical objectives for observational purposes only are as follows:

1. Patient reported and clinical outcomes.
2. Number of "failures" in each group (defined as additional surgery and/or having <12% improvement in SANE score from baseline).

ELIGIBILITY:
Inclusion Criteria:

* 70 years of age or older
* clinical and radiological diagnosis of a full thickness supraspinatus (or larger) RC tear >2cm or more than 1 full tendon
* ongoing symptoms after 3 months of physiotherapy
* a tendon amenable to partial or complete repair (as determined by pre-operative MRI)
* absence glenohumeral arthritis (Hamada < 3)
* absence of neoplastic diseases at treated site

Exclusion Criteria:

* previous surgery or pseudoparalysis on study shoulder
* complete subscapularis deficiency
* external rotation lag signs
* avascular necrosis
* post-infectious arthritis
* proximal humerus fracture
* inflammatory arithritis
* axillary nerve palsy
* concomitant tendon transfer
* neuromuscular disorder
* unable to speak/read English

Intra-operative Exclusion:

-tendon is NOT amenable to partial or complete repair

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Study feasibility - randomized | 1 year
  Percentage of patients randomized
Study feasibility - recruitment | 1 year
  Number of screened patients and proportion that are deemed eligible that consent
Study feasibility - surgery | 1 year
  Consensus among surgeon co-investigators regarding the standardized peri-operative orders and surgical techniques.

SECONDARY OUTCOMES:
ASES Score | Baseline, pre-operative
  The ASES is a patient-reported upper extremity-specific functional assessment tool and is scored out of a maximum 100 points, where 100 represents maximum function and no pain (Richards et al., 1994). It has a pain component measured on a visual analog scale as well as ten Likert-scale questions on function (e.g., put on a coat, sleep on affected side). The ASES is reliable and is validated for this population and is one of the most commonly used shoulder outcomes in North America.
ASES Score | 3 Months, post-operative
  The ASES is a patient-reported upper extremity-specific functional assessment tool and is scored out of a maximum 100 points, where 100 represents maximum function and no pain (Richards et al., 1994). It has a pain component measured on a visual analog scale as well as ten Likert-scale questions on function (e.g., put on a coat, sleep on affected side). The ASES is reliable and is validated for this population and is one of the most commonly used shoulder outcomes in North America
ASES Score | 6 Months, post-operative
  The ASES is a patient-reported upper extremity-specific functional assessment tool and is scored out of a maximum 100 points, where 100 represents maximum function and no pain (Richards et al., 1994). It has a pain component measured on a visual analog scale as well as ten Likert-scale questions on function (e.g., put on a coat, sleep on affected side). The ASES is reliable and is validated for this population and is one of the most commonly used shoulder outcomes in North America
ASES Score | 12 Months, post-operative
  The ASES is a patient-reported upper extremity-specific functional assessment tool and is scored out of a maximum 100 points, where 100 represents maximum function and no pain (Richards et al., 1994). It has a pain component measured on a visual analog scale as well as ten Likert-scale questions on function (e.g., put on a coat, sleep on affected side). The ASES is reliable and is validated for this population and is one of the most commonly used shoulder outcomes in North America
ASES Score | 24 Months, post-operative
  The ASES is a patient-reported upper extremity-specific functional assessment tool and is scored out of a maximum 100 points, where 100 represents maximum function and no pain (Richards et al., 1994). It has a pain component measured on a visual analog scale as well as ten Likert-scale questions on function (e.g., put on a coat, sleep on affected side). The ASES is reliable and is validated for this population and is one of the most commonly used shoulder outcomes in North America
EQ5D-3L | Baseline, pre-operative
  The EQ-5D is valid, reliable, responsive PROM used to document overall wellness based on 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression (Herdman et al., 2011). A single value is calculated (the value index), which indicates how good or bad a patient's health state is relative to a specified population. There are two components, VAS for general health, with 0 minimum and 100 maximum, with higher scores being more positive. The second component is a 25 point scale with minimum 5 and maximum 25 wit h lower scores more positive.
EQ5D-3L | 3 Months, post-operative
  The EQ-5D is valid, reliable, responsive PROM used to document overall wellness based on 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression (Herdman et al., 2011). A single value is calculated (the value index), which indicates how good or bad a patient's health state is relative to a specified population. There are two components, VAS for general health, with 0 minimum and 100 maximum, with higher scores being more positive. The second component is a 25 point scale with minimum 5 and maximum 25 wit h lower scores more positive.
EQ5D-3L | 6 Months, post-operative
  The EQ-5D is valid, reliable, responsive PROM used to document overall wellness based on 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression (Herdman et al., 2011). A single value is calculated (the value index), which indicates how good or bad a patient's health state is relative to a specified population. There are two components, VAS for general health, with 0 minimum and 100 maximum, with higher scores being more positive. The second component is a 25 point scale with minimum 5 and maximum 25 wit h lower scores more positive.
EQ5D-3L | 12 Months, post-operative
  The EQ-5D is valid, reliable, responsive PROM used to document overall wellness based on 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression (Herdman et al., 2011). A single value is calculated (the value index), which indicates how good or bad a patient's health state is relative to a specified population. There are two components, VAS for general health, with 0 minimum and 100 maximum, with higher scores being more positive. The second component is a 25 point scale with minimum 5 and maximum 25 wit h lower scores more positive.
EQ5D-3L | 24 Months, post-operative
  The EQ-5D is valid, reliable, responsive PROM used to document overall wellness based on 5 dimensions: mobility, self-care, usual activities, pain, anxiety/depression (Herdman et al., 2011). A single value is calculated (the value index), which indicates how good or bad a patient's health state is relative to a specified population. There are two components, VAS for general health, with 0 minimum and 100 maximum, with higher scores being more positive. The second component is a 25 point scale with minimum 5 and maximum 25 wit h lower scores more positive.
SANE Score | Baseline, pre-operative
  The Single Assessment Numeric Evaluation (SANE) score is a single question that asks patients to rate their affected shoulder as a percentage of normal to provide a simple and efficient measure of patient outcome (Gowd et al., 2019). Patients will be asked the following question: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
SANE Score | 3 Months, post-operative
  The Single Assessment Numeric Evaluation (SANE) score is a single question that asks patients to rate their affected shoulder as a percentage of normal to provide a simple and efficient measure of patient outcome (Gowd et al., 2019). Patients will be asked the following question: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
SANE Score | 6 Months, post-operative
  The Single Assessment Numeric Evaluation (SANE) score is a single question that asks patients to rate their affected shoulder as a percentage of normal to provide a simple and efficient measure of patient outcome (Gowd et al., 2019). Patients will be asked the following question: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
SANE Score | 12 Months, post-operative
  The Single Assessment Numeric Evaluation (SANE) score is a single question that asks patients to rate their affected shoulder as a percentage of normal to provide a simple and efficient measure of patient outcome (Gowd et al., 2019). Patients will be asked the following question: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
SANE Score | 24 Months, post-operative
  The Single Assessment Numeric Evaluation (SANE) score is a single question that asks patients to rate their affected shoulder as a percentage of normal to provide a simple and efficient measure of patient outcome (Gowd et al., 2019). Patients will be asked the following question: "How would you rate your affected shoulder today as a percentage of normal (0% to 100% scale with 100% being normal)?"
Constant Score | Baseline, pre-operative
  The Constant Score is validated and reliable PROM/clinical tool used to evaluate overall shoulder function based on pain, activities of daily living, and the clinical evaluation of ROM and strength (Constant & Murley, 1987). This score is widely reported in European-based literature. Minimum value is 0 and maximum value is 100, with higher scores being a better outcome.
Constant Score | 3 Months, post-operative
  The Constant Score is validated and reliable PROM/clinical tool used to evaluate overall shoulder function based on pain, activities of daily living, and the clinical evaluation of ROM and strength (Constant & Murley, 1987). This score is widely reported in European-based literature. Minimum value is 0 and maximum value is 100, with higher scores being a better outcome.
Constant Score | 6 Months, post-operative
  The Constant Score is validated and reliable PROM/clinical tool used to evaluate overall shoulder function based on pain, activities of daily living, and the clinical evaluation of ROM and strength (Constant & Murley, 1987). This score is widely reported in European-based literature. Minimum value is 0 and maximum value is 100, with higher scores being a better outcome.
Constant Score | 12 Months, post-operative
  The Constant Score is validated and reliable PROM/clinical tool used to evaluate overall shoulder function based on pain, activities of daily living, and the clinical evaluation of ROM and strength (Constant & Murley, 1987). This score is widely reported in European-based literature. Minimum value is 0 and maximum value is 100, with higher scores being a better outcome.
Constant Score | 24 Months, post-operative
  The Constant Score is validated and reliable PROM/clinical tool used to evaluate overall shoulder function based on pain, activities of daily living, and the clinical evaluation of ROM and strength (Constant & Murley, 1987). This score is widely reported in European-based literature. Minimum value is 0 and maximum value is 100, with higher scores being a better outcome.
Range of Motion | Baseline, pre-operative
  For both shoulders, forward flexion and external rotation at 0 and 90 degrees abduction will be measured with a goniometer and reported in degrees.
Range of Motion | 3 Months, post-oeprative
  For both shoulders, forward flexion and external rotation at 0 and 90 degrees abduction will be measured with a goniometer and reported in degrees.
Range of Motion | 6 Months, post-operative
  For both shoulders, forward flexion and external rotation at 0 and 90 degrees abduction will be measured with a goniometer and reported in degrees.
Range of Motion | 12 Months, post-operative
  For both shoulders, forward flexion and external rotation at 0 and 90 degrees abduction will be measured with a goniometer and reported in degrees.
Range of Motion | 24 Months, post-oeprative
  For both shoulders, forward flexion and external rotation at 0 and 90 degrees abduction will be measured with a goniometer and reported in degrees.
Isometric Strength | Baseline, pre-operative
  Measured using a hand-held dynamometer, in flexion, abduction, and external rotation.
Isometric Strength | 3 Months, post-operative
  Measured using a hand-held dynamometer, in flexion, abduction, and external rotation.
Isometric Strength | 6 Months, post-operative
  Measured using a hand-held dynamometer, in flexion, abduction, and external rotation.
Isometric Strength | 12 Months, post-operative
  Measured using a hand-held dynamometer, in flexion, abduction, and external rotation.
Isometric Strength | 24 Months, post-operative
  Measured using a hand-held dynamometer, in flexion, abduction, and external rotation.

CONTACTS AND LOCATIONS:
Overall Officials: Jarret Woodmass, MD, Principal Investigator — Pan Am Clinic